CLINICAL TRIAL: NCT01562639
Title: Nexium Capsules Specific Clinical Experience Investigation for Maintenance Therapy for Repeatedly Recurring/Relapsing Reflux Oesophagitis
Brief Title: Nexium Capsules RE Maintenance Specific Clinical Experience Investigation
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D961HC00013
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Repeatedly Recurring Esophagitis; Relapsing Reflux Esophagitis
Keywords: maintenance therapy,; repeatedly recurring,; relapsing reflux oesophagitis,; Nexium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Nexium

SUMMARY:
The purpose of this study is to collect following data in patients given Nexium capsule (Nexium) in usual post-marketing use as the maintenance therapy for repeatedly recurring/relapsing reflux oesophagitis.

DETAILED DESCRIPTION:
Nexium capsules Specific Clinical Experience Investigation for Maintenance Therapy for Repeatedly Recurring/Relapsing Reflux Oesophagitis

ELIGIBILITY:
Inclusion Criteria:

* Patients with repeatedly recurring/relapsing reflux oesophagitis who will be given Nexium for the first time as a maintenance therapy.

Exclusion Criteria:

* Patients having reflux oesophagitis when Nexium is started (Grade A, Grade B, Grade C or Grade D of Los Angeles Classification (Hoshihara's modification) on endoscopy)
* Patients having previous history of maintenance therapy for repeatedly recurring/ relapsing reflux oesophagitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with repeatedly recurring/relapsing reflux oesophagitis who will be given Nexium for the first time as a maintenance therapy.
  (Patients who had been given Nexium for the initial treatment for reflux oesophagitis can be enrolled to this investigation).
Sampling Method: Non-Probability Sample
Enrollment: 647 (Actual)
Dates: Start 2012-04; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Drug Reactions | 6 Month
  Adverse event incidence

SECONDARY OUTCOMES:
Non-recurrence rate of reflux oesophagitis | 6 Month

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Yoshida, MD, Study Director — AstraZeneca
Locations (46):
- Japan (46):
  - Research Site, Aichi
  - Research Site, Akita
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Ehime
  - Research Site, Fukui
  - Research Site, Fukuoka
  - Research Site, Fukushima
  - Research Site, Gifu
  - Research Site, Gunma
  - Research Site, Hiroshima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Ibaraki
  - Research Site, Ishikawa
  - Research Site, Kagawa
  - Research Site, Kagoshima
  - Research Site, Kanagawa
  - Research Site, Kochi
  - Research Site, Kumamoto
  - Research Site, Kyoto
  - Research Site, Mie
  - Research Site, Miyagi
  - Research Site, Miyazaki
  - Research Site, Nagano
  - Research Site, Nara
  - Research Site, Niigata
  - Research Site, Numakunai
  - Research Site, Okayama
  - Research Site, Okinawa
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Saga
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Shimane
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokushima
  - Research Site, Tokyo
  - Research Site, Tottori
  - Research Site, Toyama
  - Research Site, Wakayama
  - Research Site, Yamagata
  - Research Site, Yamaguchi
  - Research Site, Yamanashi